CLINICAL TRIAL: NCT04908254
Title: A Multi-center Randomized Control Cross-over Study to Evaluate the Safety and Effectiveness of Dayspring Active Wearable Compression Device vs. an Advanced Pneumatic Compression Device for Treating Breast Cancer Related Lymphedema
Brief Title: A Multi-center Randomized Control Cross-over Study to Evaluate the Safety and Effectiveness of the Dayspring Active Wearable Compression Device vs. an Advanced Pneumatic Compression Device for Treating Breast Cancer Related Lymphedema
Acronym: NILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KCT003
Record Dates: First submitted 2021-05-12; First posted 2021-06-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2021-05

CONDITIONS: Lymphedema; Lymphedema of Upper Arm; Lymphedema, Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Single Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dayspring Active Wearable Compression Device (Experimental): The Dayspring Active Wearable Compression Device is an FDA cleared calibrated active gradient pressure full-arm compression garment that is segmental and programmable and applies controlled sequential pressure from the distal to proximal-end of the limb in a cyclic manner.
  Interventions: Device: Crossover Device (PCD or Dayspring - alternate to first group)
- Advanced Pneumatic Compression Device (Active Comparator): A commercially available advanced pneumatic compression device that is FDA-cleared for the same indication for use as the Dayspring Wearable Compression Device.
  Interventions: Device: Crossover Device (PCD or Dayspring - alternate to first group)

INTERVENTIONS:
Device: Crossover Device (PCD or Dayspring - alternate to first group) — Cross over arms after a month of use and a month of washout period

SUMMARY:
To evaluate the Dayspring Active Wearable Compression Device in contrast to an advanced pneumatic compression device (APCD)

DETAILED DESCRIPTION:
A Multi-center Randomized Control Single Cross-over Study to Evaluate the Safety and Effectiveness of Dayspring Active Wearable Compression Device vs. an Advanced Pneumatic Compression Device for Treating Breast Cancer Related Lymphedema. To evaluate the Dayspring Active Wearable Compression Device in contrast to an advanced pneumatic compression device (APCD) in a multi-centered setting to evaluate volume, quality of life, safety, adherence, and preference.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have a diagnosis of primary or secondary unilateral upper extremity edema

Exclusion Criteria:

* Individuals with a history or presence of a systemic disorder or condition that could place the subject at increased risk from sequential compression therapy
* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Subjects with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
* Subjects must not have any diagnosed cognitive or physical impairment that would interfere with use of the device
* Diagnosis of lipedema
* Diagnosis of active or recurrent cancer (< 3 months since completion of chemotherapy, radiation therapy or primary surgery for the cancer)
* Diagnosis of Acute infection (in the last four weeks)
* Diagnosis of acute thrombophlebitis (in last 6 months)
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled)
* Diagnosis of chronic kidney disease with renal failure
* Diagnosis of epilepsy
* Subjects with poorly controlled asthma
* Any condition where increased venous and lymphatic return is undesirable
* Women who are pregnant, planning a pregnancy or nursing at study entry
* Participation in any clinical trial of an investigational substance or device during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Arm Volume Maintenance or Improvement | 1 month
  Limb volume measurement is performed by using a calibrated tape measure to measure circumference from the wrist and the ulnar styloid process and at 4cm increments to the axilla. Measurements to be taken for both upper extremities. Volume is calculated based on cylindrical segment analysis. The outcome measure is assessed as a difference or change from baseline to month 1
LYMQOL (LYMphedema Quality of Life) | 1 month
  The Lymphedema Quality of Life Questionnaire (LYMQOL), a validated disease-specific QoL tool, is also administered at baseline and month 1. Overall QoL is scored on a single item by the patient on a scale of 1-10. The outcome measure is assessed as a difference or change from baseline LYMQOL at day zero and month 1

SECONDARY OUTCOMES:
Safety/AEs | 1 month
  As assessed by reported adverse events
Therapy adherence tracking | 1 month
  A table will be provided to patient to document days of use with the device to track adherence
Patient survey on preference | 1 month
  A study survey administered at the end of the study to measure patient preference between the two devices

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - PT works, Los Altos, California
  - Ginger-K Lymphedema & Cancer Center, Morgan Hill, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rockson SG, Skoracki R. Effectiveness of a Nonpneumatic Active Compression Device in Older Adults with Breast Cancer-Related Lymphedema: A Subanalysis of a Randomized Crossover Trial. Lymphat Res Biol. 2023 Dec;21(6):581-584. doi: 10.1089/lrb.2022.0085. Epub 2023 Sep 20. PMID 37729078
- [Derived] Rockson SG, Whitworth PW, Cooper A, Kania S, Karnofel H, Nguyen M, Shadduck K, Gingerich P, Armer J. Safety and effectiveness of a novel nonpneumatic active compression device for treating breast cancer-related lymphedema: A multicenter randomized, crossover trial (NILE). J Vasc Surg Venous Lymphat Disord. 2022 Nov;10(6):1359-1366.e1. doi: 10.1016/j.jvsv.2022.06.016. Epub 2022 Aug 8. PMID 35952956